CLINICAL TRIAL: NCT06927388
Title: Myopia Progression With Freeform Open Ring Myopia Control Spectacles Versus a Commercial Peripheral Plus Myopia Control Spectacle in Chinese Children
Brief Title: Myopia Progression With Freeform Myopia Control Spectacles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRTC2024-02
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-04

CONDITIONS: Myopia, Progressive
Keywords: Myopia progression; open ring myopia control spectacle lens
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized clinical trial. There will be a total of 180 participants randomized into three groups, Group 1 - 60 participants will wear the commercial peripheral plus myopia control lens (CML).
  Group 2 - 60 participants will wear the Open Ring 1 (OR1) lens design. Group 3 - 60 participants will wear the Open Ring 2 (OR2) lens design. For each group, an equal balance of gender will be recruited and 50% of children will be aged between 6- 9 years old and 50% aged 10-12 years old.
  All groups will be required to wear spectacles for all waking hours for 12 months. After 12 months, the control group participants wearing CML will be randomised to wear either OR1 or OR2 lens designs; the Group 2 participants will continue wearing the OR1 lens for a further 12 months. The Group 3 participants will wear OR2 or OR3 (a modified design of OR2) based on their risk of myopia progression for a further 12 months.
Who Masked: Participant
Masking Description: The Investigator will not have access to this randomisation code until the trial is completed and final data analysis performed. The randomisation code for spectacles will be applied (and broken if required) by a study clinical coordinator, and clearly documented. The clinical coordinator and dispenser will not be masked from the study products. The study team will ensure that study participants are masked from the study products.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1：wear the commercial peripheral plus myopia control lens (CML). (Active Comparator): 60 participants will wear the commercial peripheral plus myopia control lens (CML) in the first year. CML will be randomised to wear either OR1 or OR2 lens designs at the second year.
  Interventions: Device: Commercial myopia control spectacle lens (CML)
- Group 2 wear the Open Ring 1 (OR1) lens (Experimental): 60 participants will wear the OR1 lens design for two years.
  Interventions: Device: freeform myopia control spectacles
- Group 3 wear the Open Ring 2 (OR2) lens (Experimental): 60 participants will wear the OR2 lens design in the first year and wear OR2 or OR3 (a modified design of OR2) based on their risk of myopia progression for a further 12 months.
  Interventions: Device: freeform myopia control spectacles

INTERVENTIONS:
Device: freeform myopia control spectacles — The open ring freeform myopia control spectacle lens designs incorporate positively powered cylindrical annular refractive elements (CARE) on the back surface with a superiorly positioned opening in each CARE. The CARE provides an effective optical myopic defocus signal for myopia control and the ring opening facilitates a defocus free zone to aid a smoother visual free transition from downgaze through to upgaze (far) vision for the wearer. The OR designs provide a difference in area and strength of myopia defocus by altering design parameters i.e. zone widths and zone powers. The OR2 and OR3 designs have wider zones and/or higher zone powers than OR1.
  Arms: Group 2 wear the Open Ring 1 (OR1) lens; Group 3 wear the Open Ring 2 (OR2) lens
Device: Commercial myopia control spectacle lens (CML) — Myoless freeform peripheral plus myopia control spectacle lens by IOT
  Arms: Group 1：wear the commercial peripheral plus myopia control lens (CML).

SUMMARY:
This is a prospective, randomized clinical trial. There will be a total of 180 participants randomized into three groups, Group 1 - 60 participants will wear the commercial peripheral plus myopia control lens (CML).

Group 2 - 60 participants will wear the Open Ring 1 (OR1) lens design. Group 3 - 60 participants will wear the Open Ring 2 (OR2) lens design. For each group, an equal balance of gender will be recruited and 50% of children will be aged between 6- 9 years old and 50% aged 10-12 years old.

All groups will be required to wear spectacles for all waking hours for 12 months. After 12 months, the control group participants wearing CML will be randomised to wear either OR1 or OR2 lens designs; the Group 2 participants will continue wearing the OR1 lens for a further 12 months. The Group 3 participants will wear OR2 or OR3 (a modified design of OR2) based on their risk of myopia progression for a further 12 months.

ELIGIBILITY:
Inclusion Criteria:

Participants enrolled in the trial must:

* be aged between 6 to 12 completed years (6 and 12 years inclusive), irrespective of gender.
* For each group, an equal balance of gender will be recruited and 50% of children will be aged between 6- 9 years old and 50% aged 10-12 years old.
* be cycloplegic autorefraction spherical component -0.50 D to -4.00D, cylinder no more than -1.50D
* be accompanied by parents/guardians who can read and comprehend Chinese and give informed consent as demonstrated by signing a record of informed consent.
* be willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator.
* have ocular health findings considered to be "normal".
* be correctable to at least 6/9.5 (20/30) or better in each eye with spectacles.
* be willing to wear the spectacles provided by the investigators for all waking hours.

Exclusion Criteria:

Participants enrolled in the trial must NOT have:

* a known allergy to, or a history of intolerance to tropicamide or topical anaesthetics.
* had strabismus and/or amblyopia.
* Anisometropia greater than 1.50D spherical equivalent
* had previous eye surgery (including strabismus surgery).
* any ocular, systemic or other condition or disease with possible associations with myopia or affecting refractive development e.g. Marfan syndrome, retinopathy of prematurity, diabetes.
* had any ocular injury or condition (including keratoconus and herpes keratitis) of the cornea, conjunctiva or eyelids.
* current orthoptic treatment or vision training.
* any anatomical, skin or other condition that would impact on the wearing of spectacles.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Currently enrolled in another clinical trial.
* No previous myopia management intervention or treatment within 3 months of enrolment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
myopic progression in one year | 12 months.
  The primary outcome measure of this study is myopic progression in one year. This is expressed as the change in spherical equivalent refractive state from baseline levels. Spherical equivalent refraction will be taken as the mean of the spherical equivalent refraction of five, reliable, cycloplegic autorefraction measurements on each eye. Myopia progression is also expressed as the change in axial length from baseline levels. Myopia progression is characterised by ocular anatomical changes, the most notable being increased axial length. This will be measured at 6 monthly intervals.

SECONDARY OUTCOMES:
myopia progression within myopia risk categories | 12 months.
  A secondary endpoint is myopia progression within myopia risk categories. Participants risk of progression will be assessed at baseline using variables such as axial length, central refraction, age, parental myopia, gender. Age, axial length percentiles and expected progression, based on published online calculators, will be converted to risk scores and categorised as low medium and high risk.
the wearer subjective experience | 12 months.
  Another secondary endpoint is the wearer subjective experience which is evaluated using a subjective quality of vision scale for various activities. Both a 1-10 scale (where 1 is poor and 10 is excellent) and a Likert scale will be used and data collected at each study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangui He, Shanghai, China